CLINICAL TRIAL: NCT01795989
Title: Novel Coils for Pediatric Musculoskeletal MRI
Brief Title: Use of Specially Designed Pediatric MR Coils on Clinical Scanners
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-2154
Record Dates: First submitted 2012-07-03; First posted 2013-02-21 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers; Musculoskeletal Complication
Keywords: Coil; MRI; safety; efficacy; musculoskeletal imaging; MSK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Research only musculoskeletal (MSK) MRI for healthy volunteers.
  Interventions: Device: 1.5T MRI Elbow Coil
- Clinical Efficacy: Clinically indicated musculoskeletal (MSK) MRI with sequences obtained using this pediatric elbow coil.
  Interventions: Device: 1.5T MRI Elbow Coil

INTERVENTIONS:
Device: 1.5T MRI Elbow Coil — Pediatric coil for musculoskeletal imaging at 1.5 Tesla for pediatric patients and healthy participants.

SUMMARY:
The purpose of this research study is to test the use of new Magnetic Resonance Imaging (MRI) coils. An MRI takes pictures of body parts using a large magnet and a computer. A coil is the part of the MRI system that collects data to make the MR images. The investigators have designed, developed, and built two child-sized coils to use when imaging elbows, wrists, knees, and ankles. These new coils will be better suited to fit infants through teenagers rather than the conventional coils used which were created for adults These MRI coils have not been approved by the US Food and Drug Administration (FDA) and are considered investigational devices.

DETAILED DESCRIPTION:
The safety and the clinical efficacy/equivalence of two pediatric 1.5T coils will be evaluated/demonstrated in two phases. Patient safety and image quality will be evaluated/demonstrated in Phase One by collecting images on healthy participants using a combination of the existing commercially available coils and the new coils. Clinical efficacy/equivalence will be evaluated/demonstrated in Phase Two by collecting standard MRI exams in pediatric patients. In Phase Two, the imaging data for a given patient will be collected by one of the two following scenarios : 1) the clinically ordered exams will be completed using a combination of the existing commercially available coils and new coil, with the images from each directly compared, or 2) the clinically ordered scans will be collected using one of the new coils and the images compared to historical de-identified MR exam, age and gender matched patient data (which were acquired using the existing commercially available coils). Results of Phase One will be reported to the IRB. Phase Two will not begin until the IRB has reviewed the results of Phase One and approved the commencement of Phase Two.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants:

* Male or female
* Age: Old enough to participate in an MR study without sedation (typically greater than 5-6 years old)

Pediatric Patients:

* Male or female
* Sent for elbow MR or superficial/small parts musculoskeletal MR imaging.
* Age: any age

Exclusion Criteria:

* Female participants who are pregnant or lactating (verbal pregnancy screens will be given for all females of child bearing potential prior to the MRI).
* Subjects with standard contraindications to MRI.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers and pediatric patients seen clinically in Radiology for a standard of care musculoskeletal (MSK) exam
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11-18 (Actual); Primary Completion 2014-12-29 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as measured by heating and comfort participant response. | Day 1
  Each participant will be monitored for adverse events during the MRI scan

SECONDARY OUTCOMES:
MRI Image Quality | Up to 3 weeks post MRI participant scan
  The following measures will be individually evaluated on 3-point scale: Overall image quality, Image uniformity overall, and Signal to Noise.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Emery, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States